CLINICAL TRIAL: NCT05596929
Title: Build-up Computed Assisted History Taking, Physical Examination and Diagnosis System of Emergency Patient Through Machine Learning (II)
Acronym: MLD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202110012RIND
Record Dates: First submitted 2022-10-10; First posted 2022-10-27 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2022-12

CONDITIONS: Internal Disease
Keywords: Artificial intelligence
MeSH Terms: interventions — Artificial Intelligence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- Experimental (Experimental)
  Interventions: Diagnostic Test: Artificial intelligence

INTERVENTIONS:
Diagnostic Test: Artificial intelligence — After the patients under triage classification to which randomly allocates in two groups. The group with AI intervention and the other without AI intervention.
  Arms: Experimental

SUMMARY:
In emergency department（ED）, physicians need to complete patient evaluation and management in a short time, which required different history taking, and physical examination skill in healthcare system.

Natural language processing（NLP） became easily accessible after the development of machine learning（ML）. Besides, electronic medical record（EMR） had been widely applied in healthcare systems. There are more and more tools try to capture certain information from the EMR help clinical workers handle increasing patient data and improving patient care.

However, to err is human. Physicians might omit some important signs or symptoms, or forget to write it down in the record especially in a busy emergency room. It will lead to an unfavorable outcome when there were medical legal issue or national health insurance review. The condition could be limited by a EMR supporting system. The quality of care will also improve.

The investigators are planning to analyze EMR of emergency room by NLP and machine learning. To establish the linkage between triage data, chief complaint, past history, present illness and physical examination. The investigators will try to predict the tentative diagnosis and patient disposition after the relationship being found. Thereafter, the investigators could try to predict the key element of history taking and physical examination of the patient and inform the physician when the miss happened. The investigators hope the system may improve the quality of medical recording and patient care.

ELIGIBILITY:
Inclusion Criteria:

* Over twenty years old
* Non-traumatic patient

Exclusion Criteria:

* Excluding the patients for administration reasons (issuing a medical certificate)
* Excluding the patients for non-emergency reasons like simply acupuncture, virus screening and prescription for medication.
* Excluding Patients who allocated to critical care station

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2022-12-12 (Actual); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Senior doctor appraisal | 24 hours
  Senior doctor appraisal which measured by an established questionnaire. Senior doctor will fill an expert-verified clinical note quality evaluation questionnaire after junior doctor finished patient interview and clinical note recording. The questionnaire is designed to use 5 points likert scale and higher scores mean a better outcome.

SECONDARY OUTCOMES:
Accuracy of diagnosis prediction | patient discharge from ED, up to 1 week
  The percentage of predicted diagnosis match the final diagnosis.
Rationality of diagnosis prediction | 24 hours
  Senior doctors will assess rationality of predicted diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Huang, Dr., Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No